CLINICAL TRIAL: NCT04977388
Title: Phase I/II Study of NORTHERA (DROXIDOPA) for Dysautonomia in Adult Survivors of Menkes Disease and Adults With Occipital Horn Syndrome: Double-blind Placebo-controlled Randomized Crossover Clinical Trial
Brief Title: NORTHERA (DROXIDOPA) for Dysautonomia in Adult Survivors of Menkes Disease and Occipital Horn Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stephen G. Kaler, MD (Other)
Responsible Party: Sponsor-Investigator, Stephen G. Kaler, MD, Professor, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 00001113
Record Dates: First submitted 2021-07-09; First posted 2021-07-26 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Menkes Disease; Occipital Horn Syndrome
Keywords: Dysautonomia
MeSH Terms: conditions — Menkes Kinky Hair Syndrome; Occipital horn syndrome; Autonomic Nervous System Diseases | interventions — Droxidopa

STUDY DESIGN:
Intervention Model Description: Double-blind Placebo-controlled Randomized Crossover Clinical Trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Northera™ (Droxidopa) (Treatment A) (Active Comparator): Northera (Droxidopa) (Treatment A) will be provided to adult subjects as a capsule with 100mg, 200mg, or 300mg of Northera (Droxidopa) contained within gelatin color capsules (sky blue and white, size 0) based on findings from the dose titration visit. These capsules are physically indistinguishable from the Treatment B (placebo) capsules. Frequency of administration (by mouth) will be twice daily for six weeks.
  Interventions: Drug: Droxidopa
- Placebo (Treatment B) (Placebo Comparator): Empty gelatin color capsules (sky blue and white, size 0) filled with cellulose microcrystalline and physically indistinguishable from Treatment A capsules. Frequency of administration (by mouth) will be twice daily for six weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Droxidopa — Subjects will self-administer capsules of Droxidopa by mouth twice daily for six weeks.
  Other Names: Northera
  Arms: Northera™ (Droxidopa) (Treatment A)
Other: Placebo — Subjects will self-administer capsules of placebo by mouth twice daily for six weeks.
  Arms: Placebo (Treatment B)

SUMMARY:
The purpose of this study is to evaluate whether Northera (Droxidopa) is safe and effective in young adults with Menkes disease who survived the most severe complications of their illness or adults with occipital horn syndrome (OHS), who have trouble with intermittent low blood pressure and other symptoms of dysautonomia. The outcomes and information from this study may help adult survivors of Menkes disease and individuals with OHS lead more normal day-to-day lives.

DETAILED DESCRIPTION:
This pilot clinical trial will evaluate the safety, tolerability, dosing, and preliminary efficacy of Northera (Droxidopa) treatment in young adults who survived the major neurodegenerative and neurocognitive effects of Menkes disease through early Copper Histidinate treatment. We hypothesize that Northera (Droxidopa) in Menkes disease survivors with symptoms of dysautonomia (e.g., syncope, dizziness, orthostatic hypotension, abnormal sinoatrial conduction, nocturnal bradycardia, and bowel or bladder dysfunction) from persistent deficiency of the copper-dependent enzyme, dopamine-β-hydroxylase, will be safe, and correct or improve blood neurochemical levels, raise systolic blood pressure, and produce symptomatic improvement and better overall quality of life. We will test this hypothesis in six to ten Menkes disease survivors or OHS patients in a double-blind placebo-controlled randomized crossover clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Adult persons with Menkes disease who survived beyond the expected natural history, attained independent ambulation, attend (or attended) school, and reached adulthood after early CuHis treatment for three years or adults with Occipital Horn Syndrome, who manifest clinical signs and symptoms of dysautonomia, e.g., orthostatic hypotension: specifically, a decrease in systolic or diastolic blood pressure of at least 20 or 10 mm Hg, respectively, within three minutes after standing, and/or chronic diarrhea: production of loose stools with or without increased stool frequency for more than four weeks immediately preceding enrollment.
2. History of at least thrice weekly occurrence of dizziness/feeling lightheaded while standing upright and/or thrice weekly episodes of diarrhea or an urgent need to defecate after food ingestion for more than four weeks immediately preceding enrollment.
3. Documented mutation in ATP7A.
4. Must sign and date an Informed Consent Form (ICF).
5. Age ≥ 18 years of age.
6. Ability to adhere to the prescribed oral Northera (Droxidopa) regimen.
7. Willingness to comply with all study visits and procedures.

Exclusion Criteria:

1. Pre-existing liver (e.g., hepatitis, biliary atresia, cirrhosis) or kidney disease (i.e., calculated glomerular filtration rate <30 ml/min).
2. History of hypertension, anti-hypertensive therapy, heart failure (or decreased ejection fraction), cardiac arrhythmia, or bleeding diatheses.
3. Any disease or condition that, in the opinion of the Investigator, has a high probability of precluding the subject from completing the study or where the subject cannot or will not appropriately comply with study requirements.
4. Any alpha-1 adrenoreceptor agonist, beta-blocker, DOPA decarboxylase inhibitor, midodrine, ephedrine, or any triptan medication as a concomitant medication.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-06-29 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events as assessed by CTCAE v5 tool | Six week periods of Active drug versus Placebo
  Grade 1-5 with increasing severity from 1 to 5

SECONDARY OUTCOMES:
Change in plasma catechol levels after Northera (Droxidopa) | Six week periods of active drug versus placebo
  Serial determinations of norepinephrine and dihydroxyphenylglycol
Changes in systolic blood pressure after Northera (Droxidopa) | Six week periods of active drug versus placebo
  Serial BP measurements including at-home monitoring
Changes in gastrointestinal symptoms after Northera (Droxidopa) | Six week periods of active drug versus placebo
  As reflected in the Irritable Bowel Syndrome-Diarrhea report
Changes in Time standing duration after Northera (Droxidopa) | Six week periods of active drug versus placebo
  Measured in time seconds
Changes in Up and Go test performance after Northera (Droxidopa) | Six week periods of active drug versus placebo
  Measured in time (seconds) needed to stand up from a chair, walk 3 m and return to a seated position on the chair.
Changes in 6 minute walk test performance after Northera (Droxidopa) | Six week periods of active drug versus placebo
  Measured in distance (meters) walked in 6 minutes

OTHER OUTCOMES:
Change in scores on the Orthostatic Hypotension Symptom Assessment questionnaire after Northera (Droxidopa) | Six week periods of active drug versus placebo
  Scores range from zero to 10 with 0 meaning no symptoms and 10 meaning the worst possible symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Stephen G Kaler, MD, Principal Investigator — Vagelos College of Physicians & Surgeons, Columbia University, New York, NY
Locations (1):
- Vagelos College of Physicians and Surgeons, Columbia University, New York, New York, United States